CLINICAL TRIAL: NCT03818100
Title: Neo-RT: Pre-operative Breast Intensity Modulated Radiotherapy in Patients Receiving Neo-adjuvant Hormonal Treatment for Breast Cancer - a Feasibility Study.
Brief Title: Neo-RT: A Study Investigating Whether Changing the Sequence of Treatments (Starting Radiotherapy Followed by Hormone Therapy Before Surgery) is Feasible
Acronym: Neo-RT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: Breast Cancer Now (Other); CRUK Cambridge Institute (Unknown)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Dr Charlotte Coles, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: Neo-RT
Record Dates: First submitted 2018-07-24; First posted 2019-01-28 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour tissue samples, blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Intensity modulated radiotherapy (IMRT) — Simultaneous integrated boost technique using IMRT: 48 Gray (Gy) and 40 Gy will treat tumour and breast tissue respectively, in 15 fractions over 3 weeks.
Drug: Endocrine therapy — Endocrine therapy will commence following completion of radiotherapy, and will continue for 20 weeks.
Procedure: Breast conserving surgery — Surgery carried out using local protocol following completion of endocrine therapy.

SUMMARY:
Four in 10 women diagnosed with breast cancer undergo mastectomy with or without breast reconstruction and less than half are satisfied with how they look unclothed. Breast conservation (removing the area with the lump only) can offer less extensive surgery and improved breast appearance, which can therefore increase well-being.

Intensity-modulated radiotherapy (IMRT) closely shapes the radiation beam to the cancer and is currently given after breast surgery. A new combination of IMRT followed by hormone treatment given before surgery, may increase the possibility of breast conservation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate
* Female
* Aged 18 years and older
* ECOG performance status 0-2
* Histology confirmed invasive breast cancer
* ER positive (Allred score 6-8)
* HER2 negative
* Palpable size ≥20mm
* Grade I-II (or grade III if considered not suitable for neo-adjuvant chemotherapy)
* Considered that radiotherapy will make breast conserving surgery easier
* No evidence of non-breast malignancy if treated with curative intent unless the patient has been disease free ≥5 years
* Unifocal or multifocal disease, i.e. tumour in the same quadrant and breast conserving surgery still feasible

Exclusion Criteria:

* Contraindications to breast radiotherapy or neo-adjuvant endocrine therapy
* Bilateral breast cancer
* Metastatic cancer
* Multicentric disease
* Concomitant medical/psychiatric problems preventing completion of study treatment or follow-up
* Pregnancy
* Breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with invasive breast cancer for planned treatment with neo-adjuvant endocrine therapy, where radiotherapy may make breast conserving surgery easier.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2018-03-26 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients successfully completing neo-adjuvant IMRT and endocrine treatment followed by beast surgery, as per study protocol. | 6 months
  Successful completion of IMRT is defined as:
  * Treatment received was either 48 Gy/15# or 40 Gy/15# with sequential boost
  * Treatment received was 'other', but the reason for different schedule was not due to toxicity related from the radiotherapy
  * Radiotherapy treatment was not delayed by 5 days or more
  * Radiotherapy treatment was delayed by 5 days or more, but the reason was not due to toxicity related from the radiotherapy
  Successful completion of endocrine treatment is defined as:
  * Patient received at least 80% of endocrine treatment received
  * Patient did not receive 80% of endocrine treatment, but the reason was not due to toxicity or toxicity related from radiotherapy or endocrine
  Successful surgery is defined as:
  * Planned date of surgery is not delayed
  * Planned date of surgery is delayed, but the reason was not due to toxicity or toxicity related to radiotherapy or endocrine treatment.

SECONDARY OUTCOMES:
Acute radiotherapy toxicity following IMRT, assessed by CTCAE v4.03 | 3 weeks
  Acute radiotherapy toxicity following IMRT, assessed by CTCAE v4.03
Mastectomy rate | 6 months
  Analysis will be descriptive, and in accordance to the statistical analysis plan.
Peri/post operative complications | 9 months
  Including:
  * Length of stay
  * Unplanned return to theatre (and reason)
  * Use of antibiotics for wound related issues
  * Number of clinic attendances for wound related problems
Volume of residual tumour and response to treatment | 6 months
  There will be a central review (2 readers) of all primary surgery histopathology reports for the secondary endpoint of pathological complete response (pCR). The histopathology slides from the surgical resection will be requested for central assessment of residual disease for all cases where there has not been a pCR. The variables that will be recorded include residual invasive tumour size in two dimensions, residual invasive tumour cellularity, number of lymph node metastases and size of the largest metastasis. A representative tumour tissue block will be selected and requested from the laboratory. Sections from the block will be taken for staining with ER and Ki67 to allow calculation of the histological assessment of residual tumour burden, and cores taken as per the protocol.
Late normal tissue toxicity, as assessed by: 1) clinicians | Annually for 5 years
  Clinician - post-radiotherapy questionnaire (with permission from IMPORT Trial Management Group and Dr Penny Hopwood)
Late normal tissue toxicity, as assessed by: 2) Patient Reported Outcome Measurements (PROMs) | Annually for 5 years
  Patient Reported Outcome Measure - Validated Breast-Q questionnaire
Late normal tissue toxicity, as assessed by: 2) Patient Reported Outcome Measurements (PROMs) | Annually for 5 years
  Patient Reported Outcome Measure - EORTC IL1 Modified BRECON23 PROM questionnaire.

OTHER OUTCOMES:
Exploratory research will be carried out to identify possible molecular and radiological biomarkers of response | 6 months post last patient recruited
  Exploratory investigation of potential biomarkers include:
  * ctDNA,
  * PBMCs,
  * Tumour molecular profiles,
  * Immunohistochemical/immunofluorescence markers of:
  Immune response (TILs) Tumour proliferation (Ki67, Geminin) DNA damage response and cell cycle checkpoint activation (including 53BP1, RAD51, ATM1, BRCA1, p53, p21 and p-chk-1) Tumour microenvironment (hypoxia)
  - Multiplexed single cell proteomics of both cellular suspensions (including whole blood) and intact tissues, to investigate the immune response and other novel markers
  Since the identification of new biomarkers correlating with disease activity and the efficacy or safety of treatment is rapidly evolving, the definitive list of biomarkers remains to be determined. However they will be detailed in an appropriate analysis plan prior to undertaking any sample analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte E Coles, MB ChB, MRCP, FRCR, PhD, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom